CLINICAL TRIAL: NCT02585284
Title: Effect of Age on Propofol-Bispectral Index Response Relationship Among Different Age Groups From Vicenarians to Nonagenarians. A New Logistic Model Compared With Traditional Sigmoid Emax Model
Brief Title: Effect of Age on Propofol-BIS Response
Acronym: BIS3
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Ashraf Dahaba, MD, Principle Investigator, Suez Canal University
Other Study IDs: MUGraz3
Record Dates: First submitted 2015-10-16; First posted 2015-10-23 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- vicenarian: 20 to 29 years. Five males and five females
- tricenarian: 30 to 39 years. Five males and five females
- quadragenarian: 40 to 49 years. Five males and five females
- quinquagenarian: 50 to 59 years. Five males and five females
- sexagenarian: 60 to 69 years. Five males and five females
- septuagenarian: 70 to 79 years. Five males and five females
- octogenarian: 80 to 89 years. Five males and five females
- nonagenarian: 90-99 years. Five males and five females

SUMMARY:
Recently, reports appeared of an 88-yr-old octogenarian exhibiting bispectral index (BIS) value of 46 before anaesthesia induction, and a 91-yr-old nonagenarian fully conscious at BIS value of 52 after propofol anaesthesia recovery. BIS algorithm was heuristically derived from a database of mostly "relatively fit, young healthy" volunteers. To date there are no studies precisely quantifying BIS response to propofol concentrations among different age groups

DETAILED DESCRIPTION:
Objective: Recently, reports appeared of an 88-yr-old octogenarian exhibiting bispectral index (BIS) value of 46 before anesthesia induction, and a 91-yr-old nonagenarian fully conscious at BIS value of 52 after propofol anesthesia recovery. BIS algorithm was heuristically derived from a database of mostly "relatively fit, young healthy" volunteers. To date there are no studies precisely quantifying BIS response to propofol concentrations among different age groups.

Methods: Investigators set Propofol estimated plasma concentrations (Cp) to gradually reach 3.5 microg·mL-1 over 3.5 min in 80 patients, five male and five female, divided by age decades from vicenarian (20-29 yr) to nonagenarians (90-99 yr). BIS values were fitted against Cp in our newly devised logistic model and traditional sigmoid Emax model. Raw BIS electroencephalography and measured propofol arterial samples determined whether changes are pharmacodynamic or pharmacokinetic asserted.

Propofol link to FDA site at FDA's Drugs@FDA web site. https://www.accessdata.fda.gov/scripts/cder/drugsatfda: http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

ELIGIBILITY:
Inclusion Criteria:

80 patients, five male and five female, divided by age decades from vicenarian (20-29 yr) to nonagenarians (90-99 yr)

Exclusion Criteria:

Patients with liver disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients, five male and five female, divided by age decades from vicenarian (20-29 yr) to nonagenarians (90-99 yr)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Difference in Bispectral Index value-TCI response curves | During Induction 3.5 minutes
  Gradual Induction with propofol over 3.5 minutes from 0 to 3.5 microgram ml-1

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyang Xiao, Study Director — Guest Professor
Locations (1):
- Ashraf Dahaba, Xi'an, China

REFERENCES:
- [Background] Schultz A, Grouven U, Zander I, Beger FA, Siedenberg M, Schultz B. Age-related effects in the EEG during propofol anaesthesia. Acta Anaesthesiol Scand. 2004 Jan;48(1):27-34. doi: 10.1111/j.1399-6576.2004.00258.x. PMID 14674970
- [Background] Dahaba AA. Different conditions that could result in the bispectral index indicating an incorrect hypnotic state. Anesth Analg. 2005 Sep;101(3):765-773. doi: 10.1213/01.ane.0000167269.62966.af. PMID 16115989
- [Background] Dahaba AA, Worm HC, Zhu SM, Bao FP, Salah A, Zakaria S, Bornemann H, Stadlbauer V, Rehak PH, Metzler H, Stauber RE. Sensitivity and specificity of bispectral index for classification of overt hepatic encephalopathy: a multicentre, observer blinded, validation study. Gut. 2008 Jan;57(1):77-83. doi: 10.1136/gut.2007.129130. Epub 2007 Aug 14. PMID 17698861
- [Background] Schnider TW, Minto CF, Shafer SL, Gambus PL, Andresen C, Goodale DB, Youngs EJ. The influence of age on propofol pharmacodynamics. Anesthesiology. 1999 Jun;90(6):1502-16. doi: 10.1097/00000542-199906000-00003. PMID 10360845
- [Derived] Dahaba AA, Xiao Z, Zhu X, Dong H, Xiong L, Rehak P, Zelzer S, Wang K, Reibnegger G. Age progression from vicenarians (20-29 year) to nonagenarians (90-99 year) among a population pharmacokinetic/pharmacodynamic (PopPk-PD) covariate analysis of propofol-bispectral index (BIS) electroencephalography. J Pharmacokinet Pharmacodyn. 2020 Apr;47(2):145-161. doi: 10.1007/s10928-020-09678-0. Epub 2020 Feb 25. PMID 32100175